CLINICAL TRIAL: NCT00260936
Title: Prevalence of Morphologic and Metabolic Anormalities in HIV Infected and Uninfected Young Men
Brief Title: Metabolic Abnormalities - HIV Infected and Uninfected Males
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: ATN 021b
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Adolescent Males; HIV positive; Treatment Naive; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HIV-negative: HIV-infected and -uninfected males, ages 12 to 24 years, of Tanner Stage 4 or 5
- HIV-positive, has never been on ART: HIV-positive, has never been on ART
- HIV-positive, non PI containing NNRTI-based regimen: HIV-positive, currently on a non-PI-containing NNRTI-based regimen for at least 12 weeks. Must never have received a total of more than 6 months of PI-containing regimen, and at least one year must have passed since receipt of last PI-containing regimen
- HIV-positive, non-NNRTI-containing PI-based regimen: HIV-positive, currently on a non-NNRTI-containing PI-based regimen for at least 12 weeks. Must never have received a total of more than 6 months of NNRTI-containing regimen, and at least one year must have passed since receipt of last NNRTI-containing regimen.

SUMMARY:
To assess whether there exist significant differences in glucose metabolism, lipids, lactate, body composition, and bone density between HIV-infected and uninfected young men.

DETAILED DESCRIPTION:
The study involves a one-time collection of health and medical history data, blood and urine specimens, and physical assessments. This study will elucidate the need for a further in-depth study to understand the pathophysiological effects of protease inhibitor (PI)-based and non-nucleoside analogue reverse transcriptase inhibitor (NNRTI)-based therapies in young men.

ELIGIBILITY:
Inclusion Criteria:

* Males age 12 years and 0 days through 24 years and 364 days.
* Tanner stage 4 or 5.
* Accessible medical history and medications history.
* Willingness to fast and complete all clinical evaluations and specimen collection.
* Willingness and ability to give informed consent or assent with parental/legal guardian permission, where required.

Group 1: HIV-Negative Control Subject Specific Inclusion Criteria

* All subjects for Group 1 will be tested for HIV-1 to confirm negativity unless they have a documented negative antibody test within the last three months of study entry.
* Willingness and ability to give informed consent for HIV testing. Groups 2, 3, and 4: HIV-Positive Subject Specific Inclusion Criteria
* HIV-1 infection as documented by a positive result on any of the following licensed tests at any time: any antibody test confirmed by Western blot, HIV culture, plasma HIV-1 RNA PCR >1,000 copies/ml or HIV-1 DNA PCR.
* Horizontal HIV infection transmission (non-perinatal, non-transfusion acquired infection).
* Group 2: Currently not on ART and must never have received ART.
* Group 3: Currently on a NNRTI, non-PI containing regimen for three or more months, must never have received a total of more than six months of PI-containing regimen and at least one year must have passed since receipt of last PI-containing regimen.
* Group 4: Currently on a PI, non-NNRTI containing regimen for three or more months, must never have received a total of more than six months of NNRTI-containing regimen and at least one year must have passed since receipt of last NNRTI-containing regimen.

Exclusion Criteria:

* Transgender male to female (MTF) or female to male (FTM) youth
* Refusal to fast for the 8 hours before collection of laboratory specimen requiring fasting.
* Unable to obtain medical/medications history.
* History of anorexia or bulimia.
* Type I Diabetes Mellitus.
* Type II Diabetes Mellitus and cannot omit diabetes medication for the 48-hour period prior to laboratory specimen collection for oral glucose tolerance test (OGTT).
* Current use or use within the past 6 months of oxandrolone, nandrolone, oxymetholone, stanozolol, or any other synthetic anabolic/androgenic agents.
* Current use or use within the past 6 months of pharmacologic doses of growth hormone. Physiologic growth hormone replacement therapy is permitted, as long as dosages meet the following specifications:
* Adolescents in puberty - less than or equal to an equivalent of 0.1 mg/kg/day
* Adolescents past puberty - less than or equal to an equivalent of 0.025 mg/kg/day
* Current use or use within the past 6 months of pharmacologic doses of testosterone. Physiologic testosterone replacement therapy is permitted as long as dosages meet the following specifications:
* Injection - no more than 400 mg/month of testosterone enanthate
* Patch - no more than 5 mg/day (e.g. Testoderm, Androderm)
* Gel in pre-packaged doses - no more than 7.5 g/day of gel (e.g. Androgel, Testim)

Ages: 12 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Approximately 250 subjects will be enrolled in the study. The number of subjects enrolled in each study group will be as follows: 50 HIV-negative subjects; 100 HIV-positive subjects who are antiretroviral therapy (ART) naïve; and two groups of up to 50 HIV-positive subjects each, one on an NNRTI-based regimen and the other on a PI-based regimen.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Aldrovandi, MD, Study Chair — Children's Hospital Los Angeles
Locations (13):
- United States (12):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Childrens Hopital National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnoistic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Children's Hopsital of Boston, Boston, Massachusetts
  - Mount Siani Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org